CLINICAL TRIAL: NCT06873828
Title: Evaluation of the Efficacy and Safety of Wearable ECG (AT-Patch) in Patients With Hypertrophic Cardiomyopathy Requiring 48-Hour Holter Monitoring : A Prospective Superiority Study
Brief Title: Evaluation of the Efficacy and Safety of Wearable ECG (AT-Patch) in Patients With Hypertrophic Cardiomyopathy Requiring 48-Hour Holter MonitoringEvaluation of the Efficacy and Safety of Wearable ECG (AT-Patch) in Patients With Hypertrophic Cardiomyopathy Requiring 48-Hour Holter Monitoring
Acronym: ATP-HCM
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024-3479-001
Record Dates: First submitted 2025-02-26; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Hypertrophic Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: ATP-C135 — A wearable long-term electrocardiogram monitoring device that monitors electrocardiograms by attaching it for up to 14 days.
Device: ATP-C75 — A wearable long-term electrocardiogram monitoring device that monitors electrocardiograms by attaching it for up to 7 days.

SUMMARY:
* Validation of validity, superiority, and safety of data analysis results using AT-Patch compared to 48-hour Holter test results
* Number of subjects: 100 (including 10% dropout rate)
* Performance and safety were verified by simultaneously attaching a 48-hour Holter and a wearable Holter device (ATP-C75 or ATP-C135).

DETAILED DESCRIPTION:
Prospective, sequential, superiority test Patients diagnosed with hypertrophic cardiomyopathy who require 48-hour Holter monitoring.

* 48-hour Holter vs ATP-C75 (48-hour comparison/total time comparison)
* 48-hour Holter vs ATP-C135 (48-hour comparison/total time comparison)
* Comparison between IDs

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects aged 19 years or older
2. Subjects diagnosed with hypertrophic cardiomyopathy who require 48-hour Holter examination

Exclusion Criteria:

1. Those judged by the investigator to be unsuitable for this clinical trial or those who may increase the risk due to participation in the clinical trial
2. Those with sensitive or allergic skin, skin diseases such as skin cancer or rashes
3. Those with pacemakers, implantable cardioverter-defibrillators, or other implantable electrical devices
4. Pregnant women

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Comparison of arrhythmia detection rates between the test group and the control group after using a medical device for clinical trials | ATP-C75 : 7day , ATP-C135 : 14day
  * 48-hour Holter vs ATP-C75 (48-hour comparison/7days)
  * 48-hour Holter vs ATP-C135 (48-hour comparison/14days)

SECONDARY OUTCOMES:
Arrhythmia detection rate by test time in the test group and control group after using the clinical trial medical device | ■48-hour Holter vs ATP-C75 (48-hour comparison/7days) ■48-hour Holter vs ATP-C135 (48-hour comparison/ 14days)
  Comparison of control and test period (48hrs vs total time) Comparison by disease type Comparison of test period ATP-C135 : 14day / No f/u
  ■ Safety Issue ATP-C75 : 7day ATP-C135 : 14day
Comparison of the concordance rate of the analysis results of the simultaneous attachment time in the test group and control group after using the clinical trial medical device | ■48-hour Holter vs ATP-C75 (48-hour comparison) ■48-hour Holter vs ATP-C135 (48-hour comparison)
  Comparison of control and test period (48hrs vs total time) Comparison by disease type Comparison of test period ATP-C135 : 14day / No f/u
  ■ Safety Issue ATP-C75 : 7day ATP-C135 : 14day
User response evaluation (satisfaction) in the test group and control group after using the clinical trial medical device | ■48-hour Holter : 48hrs ■ATP-C75 : 7days ■ATP-C135 : 14days
  Comparison of control and test period (48hrs vs total time) Comparison by disease type Comparison of test period ATP-C135 : 14day / No f/u
  ■ Safety Issue ATP-C75 : 7day ATP-C135 : 14day
Arrhythmia detection rate in the test group and control group by hypertrophic cardiomyopathy subtype (Apical HCM, Non-apical HCM) | ■48-hour Holter vs ATP-C75 (48-hour comparison/7days) ■48-hour Holter vs ATP-C135 (48-hour comparison/ 14days)
  Comparison of control and test period (48hrs vs total time) Comparison by disease type Comparison of test period ATP-C135 : 14day / No f/u
  ■ Safety Issue ATP-C75 : 7day ATP-C135 : 14day
Arrhythmia detection rate by test group (ATP-C75, ATP-C135) | ■ATP-C75 vs ATP-C135 ( 7days vs 14days )
  Comparison of control and test period (48hrs vs total time) Comparison by disease type Comparison of test period

IPD SHARING:
Plan to Share IPD: No
The individual data of the subjects will be pseudonymized/anonymized in accordance with ICH GCP and recorded in the case record sheet, and only the participating researchers will be able to access the data. Monitoring will be conducted by a monitor designated by the client to conduct SDV, and the CRF for which SDV has been completed will be collected at the end of the study with the signature of the PI.

REFERENCES:
- [Background] Rowin EJ, Das G, Madias C, Hsu M, Crosson L, Turakhia MP, Maron BJ, Maron MS. Extended ambulatory ECG monitoring enhances identification of higher-risk ventricular tachyarrhythmias in patients with hypertrophic cardiomyopathy. Heart Rhythm. 2025 Jul;22(7):1696-1704. doi: 10.1016/j.hrthm.2024.09.040. Epub 2024 Sep 20. PMID 39307380
- [Background] Weissler-Snir A, Chan RH, Adler A, Care M, Chauhan V, Gollob MH, Ziv-Baran T, Fourey D, Hindieh W, Rakowski H, Spears DA. Usefulness of 14-Day Holter for Detection of Nonsustained Ventricular Tachycardia in Patients With Hypertrophic Cardiomyopathy. Am J Cardiol. 2016 Oct 15;118(8):1258-1263. doi: 10.1016/j.amjcard.2016.07.043. Epub 2016 Jul 29. PMID 27567133
- [Background] Bansal A, Joshi R. Portable out-of-hospital electrocardiography: A review of current technologies. J Arrhythm. 2018 Feb 23;34(2):129-138. doi: 10.1002/joa3.12035. eCollection 2018 Apr. PMID 29657588